CLINICAL TRIAL: NCT01134237
Title: Intrapleural Thrombolytic Treatment With Urokinase for Retained Hemothorax: A Prospective Double-blinded Randomized Multicenter Study
Brief Title: Intrapleural Urokinase for Retained Hemothorax
Acronym: NTUH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chin-Chih Chang, Department of Traumatology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200908047M; NTUH. 99-N1457 (Other Grant/Funding Number: National Taiwan University Hospital)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Retained Hemothorax
Keywords: non-surgical rate
MeSH Terms: interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urokinase (Active Comparator): arm of interest
  Interventions: Drug: urokinase
- Control (Placebo Comparator): Normal saline as a placebo for control arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: urokinase — intrapleural urokinase injection
  Arms: Urokinase
Drug: placebo — Normal saline as a placebo for control arm
  Arms: Control

SUMMARY:
Intrapleural thrombolytic treatment with urokinase for retained hemothorax is effective and safe. However, previous study was limited in prospective observation study without control group.

DETAILED DESCRIPTION:
We will recruit 32 patients in this study. The patients with retained hemothorax will be randomly divided into the urokinase group and the placebo group. In the urokinase group, urokinase 100,000 IU in 100 mL NaCl will be injected into the intrapleural space. We will record the daily drainage amount and evaluate the therapeutic effect by the chest X-ray. The therapeutic effect, safety, hospital stay, and medical cost between the two groups will be compared. This study will be done in four medical centers in northern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Retained hemothorax: it is defined as chest X-ray revealing obvious blood clot in pleural cavity after tube thoracostomy drainage for 3 days. The chest tubes are in good location and have no obstruction. The physician thinks the blood clot is difficult to drain.
2. Age: full 18 year-old

Exclusion Criteria:

1. Pregnancy
2. Active bleeding
3. Coagulopathy, e.g. congenital or acquired coagulation abnormality, platelet count less than 100,000 /μL, international normalized ratio (INR) more than 1.5, or partial thromboplastin time, PTT, more than 50 seconds after treatment.
4. Cerebrovascular accident within 30 days
5. History of intracranial tumor or vascular abnormality
6. Have received thoracic surgery
7. Have received pleurodesis
8. Wish to receive thoracoscopic surgery for hematoma evacuation directly
9. Allergy to urokinase
10. Sepsis
11. Shock
12. People who are less than 18 years of age, prisoners, aborigines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
non-surgical rate | about 5 days
  Complete response and partial response

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chih Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Chin-Chih Chang, Taipei, Taiwan, Taiwan